CLINICAL TRIAL: NCT07298642
Title: Proton Therapy in Extended-field Irradiation for Cervical Cancer
Brief Title: Extended-field Proton Therapy for Cervical Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Clinical Associate Professor, Attending Physician, Jenny Ling-Yu Chen MD PhD, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202502003RINB; TGOG7001 (Other Grant/Funding Number: Taiwanese Gynecologic Oncology Group (TGOG) study)
Record Dates: First submitted 2025-11-26; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; proton therapy; extended field
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Extended field radiation therapy (Proton vs Photon)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proton extended-field radiotherapy (Experimental): Proton extended-field radiotherapy
  Interventions: Radiation: Proton extended field radiation therapy
- Photon extended-field radiotherapy (Active Comparator): Photon extended-field radiotherapy
  Interventions: Radiation: Photon extended field radiation therapy

INTERVENTIONS:
Radiation: Proton extended field radiation therapy — Proton extended field radiation therapy
  Arms: Proton extended-field radiotherapy
Radiation: Photon extended field radiation therapy — Photon extended field radiation therapy
  Arms: Photon extended-field radiotherapy

SUMMARY:
Severe lymphopenia is a common complication of extended-field radiotherapy in cervical cancer, significantly impacting immune function and clinical outcomes. This study aims to evaluate whether proton therapy, with its superior dose distribution, can reduce lymphopenia and improve survival and toxicity profiles compared to photon therapy.

DETAILED DESCRIPTION:
This study is a prospective, observational cohort study designed to evaluate the effects of proton therapy and photon therapy in patients with stage IIIC1 or IIIC2 cervical cancer undergoing extended-field radiotherapy. Primary data collection will include clinical outcomes, radiotherapy-related toxicities, lymphocyte counts, and immune cell subsets (e.g., CD4, CD8, CD19, and CD16+56), measured at baseline, during treatment, and post-treatment. Secondary data collection will involve tissue banking for future translational research projects, including serum, plasma, and whole blood for DNA analysis.

The study will be conducted in two tertiary cancer centers (CGMH and NTUCC), with individual patient participation proton or photon treatment approximately 9 weeks, followed by an additional five years for long-term follow-up to assess survival outcomes and late toxicities. This design enables robust comparison of the therapeutic impact of proton and photon therapies on clinical and immunological endpoints, providing evidence to guide personalized treatment decisions in cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cervical cancer, stage ≥ IIIC.
* Age between 20 and 85 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Eligible for extended-field radiotherapy as determined by the treating physician.
* Induction chemotherapy with paclitaxel and carboplatin is allowed if the duration is ≤ 6 weeks or ≤ 2 cycles.
* RT alone, or concurrent single-agent chemotherapy with weekly cisplatin or carboplatin during radiation therapy is allowed, while the use of any other concurrent antineoplastic agents is prohibited.
* Consolidative chemotherapy or immunotherapy after radiation therapy is allowed.

Exclusion Criteria:

* Prior history of pelvic or abdominal radiotherapy.
* Presence of distant metastases or other active malignancies within the past 5 years, excluding non-melanoma skin cancer.
* Severe comorbid conditions, such as uncontrolled diabetes, cardiovascular disease, or autoimmune disorders, that may interfere with treatment or study participation.
* Pregnancy or breastfeeding at the time of enrollment.
* Psychiatric or social conditions that would limit compliance with study requirements or follow-up.

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Lymphocyte Counts | Baseline; Weeks 3-5 of radiotherapy; 2 weeks after radiotherapy completion
  Lymphocyte Counts: The absolute lymphocyte count will be measured pre-treatment, during treatment, and post-treatment. Severe lymphopenia is defined as an absolute lymphocyte count <500/μL
Immune Cell Subsets | Baseline; Weeks 3-5 of radiotherapy; 2 weeks after radiotherapy completion
  Immune Cell Subsets: The percentage of CD4 (%), CD8 (%), CD19 (%), and CD16+56 (%) will be monitored to assess the immune response to therapy

SECONDARY OUTCOMES:
Radiotherapy-Related Toxicities | Follow-up for five years
  * Radiotherapy-Related Toxicities: Toxicity levels will be assessed using the CTCAE grading system. Acute and late toxicities will be documented, with a focus on gastrointestinal, hematological, genitourinary, and skin toxicities as part of the comparison between proton and photon therapy.
Survival outcomes | Follow-up for five years
  * Overall Survival (OS): The time from the start of treatment to death from any cause.
  * Progression-Free Survival (PFS): The time from the start of treatment to disease progression or death, whichever occurs first. PFS provides insight into the therapeutic efficacy and disease control achieved by each treatment modality.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided